CLINICAL TRIAL: NCT03624218
Title: Prolonged Exposure Therapy (PE) for Posttraumatic Stress Disorder (PTSD) in Spinal Cord Injury (SCI): a Randomized Controlled Trial
Brief Title: Outcomes After Spinal Cord Injury (OASIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-410
Record Dates: First submitted 2018-07-25; First posted 2018-08-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Posttraumatic Stress Disorder; Spinal Cord Injuries
Keywords: PTSD; SCI; PE; Prolonged Exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Participants in the control arm will not receive the PE therapy, but they will rather receive the standard clinical treatment receive by all SCI patients at BIR. This includes an evaluation by a licensed psychologist and continued follow-up psychotherapy as needed. This therapy does not consist of trauma-focused therapy and will be summarized in the analysis as a part of standard of care. TAU participants will have a posttreatment assessment, as well as follow-up assessments at one and 6 months
- Intervention (Experimental): Participants randomized to the PE intervention will receive 2-3, 60-minute sessions each week for 4-6 weeks (12 total sessions). Treatment is manualized, and includes education about common reactions to trauma, breathing retraining, prolonged (repeated) imaginal exposure to trauma memories, repeated in vivo exposure to situations that participants are avoiding due to trauma-related fear, and discussion of thoughts and feelings related to exposure exercises.
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — Using a combination of In vivo and Imaginal exposure, Prolonged Exposure therapy aims to treat those with Posttraumatic Stress Disorder.
  Arms: Intervention

SUMMARY:
The study evaluates the effectiveness of Prolonged Exposure Therapy on a population of individuals with spinal cord injuries. Participants will be randomly assigned to either a treatment as usual or Prolonged Exposure therapy group.

DETAILED DESCRIPTION:
The National Spinal Cord Injury Statistical Center estimates 282,000 people in the US live with spinal cord injury (SCI), with approximately 17,000 new cases occurring each year. There has been tremendous progress in the medical and rehabilitative management of people who have sustained SCI including improved clinical outcomes, decreased mortality during the first year after injury, and increased life expectancy. However, there has been less innovation to support mental health among SCI patients. In addition, most attention has been focused on addressing the elevated rate of depression in people with SCI. Much less attention has focused on Posttraumatic Stress Disorder (PTSD) despite prevalence estimates suggesting that it affects up to 60% of those with SCI compared to only 7% of the general US population. Notably, PTSD prevalence estimates among those with SCI are similar to those reported in a recent meta-analysis that showed 23% of veterans who served in conflicts in Afghanistan and Iraq experienced PTSD. PTSD can be a disabling psychological consequence of surviving SCI, impacting one's health and function, including the ability to return to normal activities of daily life (e.g., work, school, social relationships). Further, PTSD is one of the most costly of all anxiety disorders because of work impairment, hospitalization, and physician visits. Fortunately, there are highly effective treatments for PTSD. The most researched and effective treatment for PTSD is Prolonged Exposure Therapy. In 12 sessions over 6 weeks, 85% of patients with PTSD respond to treatment and the dropout rate is similar to all other treatments (20%). Thus far, PE has been tested within survivors of combat, rape, non-sexual assault, motor vehicle collisions, natural disasters, males/females, civilians/military, and adolescents. However, this treatment has not been tested with this population despite evidence that there is no reason to expect it would not be effective. In summary, greater attention has focused in recent years on PTSD and developing evidence-based approaches to treat it due to the number of veterans returning from conflicts in the Middle East dealing with the condition. Despite this increased overall focus on PTSD, and despite the higher prevalence of PTSD among people with SCI than among those in the general population, the literature lacks studies of PTSD in patients with SCI. Thus, the primary aim of the current study (Field Initiated Projects Program - Research HHS-2017-ACL-NIDILRR-IFRE-0192) is to use a randomized controlled trial (RCT) to evaluate the efficacy of Prolonged Exposure Therapy (PE) on PTSD symptoms among SCI patients. First, the investigators expect that individuals with SCI who receive the PE intervention for PTSD will show statistically significantly greater improvements in PTSD symptoms relative to the treatment as usual (TAU) control group. Second, the investigators hypothesize that compared to the TAU control group, those randomized to the PE will experience: a) significantly greater reduction in pain, b) significantly greater improvement in depression, c) significantly greater improvement in sleep, and d) significantly greater improvement in quality of life. Finally, we expect that PE will be feasible and acceptable in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the trauma service at BUMC or Inpatient service at BIR
* Patients with SCI
* Patients at least 30 days post injury (to insure proper PTSD diagnosis)
* Patients ages 18 and older
* Patients who have a positive PTSD screen using PTSD Symptom Scale - Interview for DSM-5 (PSSI-5)

Exclusion Criteria:

* Patients in police custody
* Non-English speaking
* Patients with severe cognitive impairment (will be assessed through chart review and with the Cognistat)
* Patients who are acutely suicidal and/or have been admitted for a suicide attempt
* Patients who are actively psychotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
The PTSD Symptom Scale - Interview for DSM-5 (PSSI-5) | Used to assess change in Posttraumatic Stress entomology at Baseline, 6 week, 10 week, and 32 week about their past two week experiences.
  The PSSI-5 is a 24-item, semi-structured interview that assesses PTSD symptoms in the past two weeks, and makes a diagnostic determination based on the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria. The interviewer rates participant responses to symptom questions on a 5-point scale of frequency and severity, from 0 ("Not at all") to 4 ("6 or more times a week/severe") with a higher total score meaning more Posttraumatic stress symptoms.

SECONDARY OUTCOMES:
The MINI International Neuropsychiatric Interview (MINI) | Assessed at Baseline about past month and lifetime experiences.
  It assesses multiple diagnoses including Posttraumatic Stress Disorder, Major Depressive Depression, and Generalized Anxiety Disorder.
The Beck Depression Inventory-II (BDI-II) | Assessed at Baseline, at every Prolonged Therapy Session, 6 week, 10 week, and 32 week about their past month experiences.
  The BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
Post-Traumatic Cognitions Inventory (PTCI) | Assessed at Baseline, at every Prolonged Therapy Session, 6 week, 10 week, and 32 week about their past month experiences.
  The Post-Traumatic Cognitions Inventory (PTCI) is a 36-item instrument that assesses dysfunctional post-trauma cognitions across self, world, and self-blame to yield a total score. The PCTI is rated on a Likert-type scale ranging from 1 (totally disagree) to 7 (totally agree)
Numerical Rating Scale (NRS) | Assessed at Baseline,10 week, and 32 week about their past week experience.
  The Numerical Rating Scale (NRS) has been validated as a measure of pain intensity and is one of the most commonly used measures in assessing pain. The NRS asks patients to rate their pain severity on a 0 to 10 scale, with 0 being "no pain" to 10 being "so severe that you can't stand it."
Pittsburgh Sleep Quality Index Addendum for PTSD (PSQI-A) | Assessed at Baseline,10 week, and 32 week about their past month experience.
  The Pittsburgh Sleep Quality Index Addendum for PTSD (PSQI-A), is a 7-item, self-report instrument that assesses the frequency of disruptive nocturnal behaviors, which are often associated with PTSD. Each item is rated on a 0-3 scale referring to frequency of each disturbance, where 0=not in the past month, 1=less than once a week, 2=once or twice a week, and 3=three or more times a week. A global score is obtained from the sum of all seven items, and has a range of 0-21. The PSQI-A includes three additional items regarding the frequency of anxiety and anger accompanying DNB and the timing of these events during the night.
SCI Quality of Life- Positive Affect & Well-Being - Short Form (SCI-QOL) | Assessed at Baseline,10 week, and 32 week about their past week Past 7 Days experience.
  SCI Quality of Life- Positive Affect & Well-Being - Short Form (SCI-QOL) is a 10- item, self-report measure that assesses participants' positive affect and well-being (e.g., "I thought positively about my future") in the past 7 days on a Likert scale of 1-5, with 1 representing "never" and 5 representing "always."
Posttraumatic Growth Inventory (PTGI) | Assessed at 32 week about their past week Past Month experience.
  The Posttraumatic Growth Inventory (PTGI) is an instrument for assessing positive outcomes reported by persons who have experienced traumatic events. This 21-item scale includes factors of New Possibilities, Relating to Others, Personal Strength, Spiritual Change, and Appreciation of Life. A 6-point Likert response format was used, ranging from "I did not experience this change as a result of my crisis" (scored 0), to "I experienced this change to a very great degree as a result of my crisis" (scored 5). Intermediate scores were given for a very small degree (1), a small degree (2), a moderate degree (3), and a great degree (4).
Alcohol Use Disorder Identification Test-Consumption (AUDIT-C) | Assessed at Baseline,10 week, and 32 week about their past week Past Year experience.
  Alcohol Use Disorder Identification Test-Consumption (AUDIT-C) is a 3-item alcohol screen that can identify problem alcohol use. The AUDIT-C is scored o a scale of 0-12, each question has 5 answer choices with "a" being 0 points and "e" being 4 points.
Drug use | Assessed at Baseline,10 week, and 32 week about their past week Past Year experience.
  Single Items and the Drug Abuse Screening Test (DAST) is used to assess the use of specific substances.
Therapy history | Assessed at Baseline, 6 week, 10 week, and 32 week about their Recent experiences.
  Therapy history is assessed via a 5-item face valid questionnaire made for the study. Questions ask about current and recent therapy and medication use in order to account for any outside therapy the TAU or PE participants might be getting using "yes" or "no" and open-ended responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Institute for Rehabilitation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Douglas ME, Bennett M, Jones KA, Pogue JR, Chauvette GV, Sikka S, Driver S, Hamilton R, Curcio N, Patel S, Wierzchowski A, Adams M, Thomas EV, Turner E, Leonard K, Carl E, Foreman M, Warren AM, Powers MB. Prolonged exposure for posttraumatic stress disorder following spinal cord injury: A randomized controlled trial. Rehabil Psychol. 2025 Aug;70(3):240-254. doi: 10.1037/rep0000580. Epub 2024 Aug 29. PMID 39207423